CLINICAL TRIAL: NCT02131636
Title: Efficacy and Safety of AGN-199201 in Patients With Persistent Erythema Associated With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199201-004
Record Dates: First submitted 2014-05-05; First posted 2014-05-06 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Erythema; Rosacea
MeSH Terms: conditions — Erythema; Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AGN-199201 (Experimental): AGN-199201 applied to the face once daily for 29 days.
  Interventions: Drug: AGN-199201
- Vehicle (Placebo Comparator): Vehicle to AGN-199201 applied to the face once daily for 29 days.
  Interventions: Drug: Vehicle to AGN-199201

INTERVENTIONS:
Drug: AGN-199201 — AGN-199201 applied to the face once daily for 29 days.
  Arms: AGN-199201
Drug: Vehicle to AGN-199201 — Vehicle to AGN-199201 applied to the face once daily for 29 days.
  Arms: Vehicle

SUMMARY:
This study will evaluate the safety and efficacy of AGN-199201 once daily compared to vehicle for the treatment of persistent moderate to severe facial erythema associated with rosacea.

ELIGIBILITY:
Inclusion Criteria:

-Moderate to severe persistent facial erythema associated with rosacea.

Exclusion Criteria:

* Greater than 3 inflammatory lesions on the face
* Current treatment with monoamine oxidase (MAO) inhibitors
* Raynaud's syndrome, narrow angle glaucoma, orthostatic hypotension, scleroderma or Sjogren's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Lynchburg, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN-199201 | Vehicle
Started | 222 | 218
Completed | 210 | 213
Not Completed | 12 | 5
Not completed — Personal Reasons | 4 | 4
Not completed — Lost to Follow-up | 4 | 0
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-199201 | Vehicle | Total
Number analyzed (Participants) | 222 | 218 | 440
Age, Customized [Number; unit: Participants]
  18 to 64 years | 189 | 194 | 383
  >=65 years | 33 | 24 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 175 | 347
  Male | 50 | 43 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With at Least a 2-Grade Decrease From Baseline on Both Clinician Erythema Assessment (CEA) and Subject Satisfaction Assessment (SSA) 5-point Scales
Description: The investigator assessed the patient's overall severity of erythema in the treatment area on the 5 point CEA scale (ranging from 0=clear skin with no signs of erythema to 4=severe erythema/fiery redness). The patient assessed the overall severity of rosacea facial redness in the treatment area on the 5 point SSA scale (ranging from 0=no signs of unwanted redness to 4=severe redness). The percentage of patients with at least a 2 grade decrease (improvement) on both CEA and SSA from baseline was evaluated over the 12-hour evaluation period (hours 3, 6, 9, and 12) postdose on day 29. Baseline was defined as the measurement at predose on Day 1.
Time Frame: Baseline, Day 29 (Hours 3, 6, 9, and 12)
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN-199201 | Vehicle
Number analyzed (Participants) | 222 | 218
Percentage of Patients
  Day 29, Hour 3 (N=222, 216) | 11.9 | 5.5
  Day 29, Hour 6 (N=222, 216) | 15.5 | 8.3
  Day 29, Hour 9 (N=222, 216) | 17.7 | 6.0
  Day 29, Hour 12 (N=222, 216) | 14.8 | 6.0

2. Secondary Outcome: Percentage of Patients With at Least a 2-Grade Decrease From Baseline on the SSA 5-point Scale
Description: The patient assessed the overall severity of rosacea facial redness in the treatment area on the 5 point SSA scale (ranging from 0=no signs of unwanted redness to 4=severe redness). The percentage of patients with at least a 2 grade decrease (improvement) from baseline was evaluated over the 12-hour evaluation period (hours 3, 6, 9, and 12) postdose on day 29. Baseline was defined as the measurement at predose on Day 1.
Time Frame: Baseline, Day 29 (Hours 3, 6, 9, and 12)
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN-199201 | Vehicle
Number analyzed (Participants) | 222 | 218
Percentage of Patients
  Day 29, Hour 3 | 20.1 | 11.1
  Day 29, Hour 6 | 23.3 | 12.9
  Day 29, Hour 9 | 23.3 | 12.0
  Day 29, Hour 12 | 25.0 | 11.5

3. Secondary Outcome: Percent Change From Baseline in Rosacea Facial Redness as Measured by Digital Imaging Analysis (DIA)
Description: Rosacea facial redness in the treatment area was measured by DIA. The percent change was evaluated over the 12-hour evaluation period (hours 3, 6, 9, and 12) postdose on Day 29. Baseline was defined as the measurement at predose on Day 1. A negative number change from baseline indicates a decrease in facial redness (improvement), and a positive number change from baseline indicates an increase in facial redness (worsening).
Time Frame: Baseline, Day 29 (Hours 3, 6, 9, and 12)
Population: Intent-to-Treat: all randomized patients with data at the time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | AGN-199201 | Vehicle
Number analyzed (Participants) | 222 | 218
Percent Change
  Day 29, Hour 3 | -21.37 (94.693) [-100.0 to 1097.0] | 61.54 (428.943) [-100.0 to 4699.1]
  Day 29, Hour 6 | -14.22 (97.835) [-100.0 to 750.3] | 75.09 (498.844) [-99.9 to 4668.5]
  Day 29, Hour 9 | -8.00 (92.893) [-100.0 to 1127.4] | 71.18 (398.072) [-98.9 to 3723.4]
  Day 29, Hour 12 | -5.35 (98.547) [-100.0 to 1211.9] | 74.16 (415.301) [-99.4 to 4894.8]

4. Secondary Outcome: Percentage of Patients Reporting Treatment Satisfaction on the Satisfaction Assessment for Rosacea Facial Redness (SA-RFR) Questionnaire Item 9
Description: The SA-RFR questionnaire item 9 is completed by patients assessing treatment satisfaction on facial redness. Patients reporting treatment satisfaction as "very satisfied" or "satisfied" are noted. The percentage of patients was evaluated over the 12-hour evaluation period (hours 3, 6, 9, and 12) postdose on Day 29.
Time Frame: Day 29 (Hours 3, 6, 9, and 12)
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN-199201 | Vehicle
Number analyzed (Participants) | 222 | 218
Percentage of Patients
  Day 29, Hour 3 | 45.9 | 27.5
  Day 29, Hour 6 | 43.7 | 24.3
  Day 29, Hour 9 | 43.2 | 23.4
  Day 29, Hour 12 | 41.9 | 24.8

5. Secondary Outcome: Change From Baseline on the SA-RFR Questionnaire Item #4
Description: The SA-RFR questionnaire item 4 is completed by patients assessing how much their face burned due to facial redness on a 5 point scale (range 0=does not burn at all and 4=burns a lot). Patients were evaluated over the 12-hour evaluation period (hours 3, 6, 9, and 12) postdose on Day 29. A lower score change from baseline (negative number) indicates a decrease in facial redness (improvement), and a higher score change from baseline (positive number) indicates an increase in facial burning (worsening).
Time Frame: Baseline, Day 29 (Hours 3, 6, 9, and 12)
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AGN-199201 | Vehicle
Number analyzed (Participants) | 130 | 149
Scores on a Scale
  Baseline | 1.8 (0.83) | 1.9 (0.85)
  Day 29, Hour 3 | -1.5 (0.93) | -1.5 (0.95)
  Day 29, Hour 6 | -1.5 (0.91) | -1.5 (0.98)
  Day 29, Hour 9 | -1.5 (0.97) | -1.5 (0.96)
  Day 29, Hour 12 | -1.5 (0.97) | -1.5 (0.95)

6. Secondary Outcome: Percentage of Patients With at Least a 1-Grade Decrease From Baseline on the SSA 5-point Scale
Description: The patient assessed the overall severity of rosacea facial redness in the treatment area on the 5 point SSA scale (ranging from 0=no signs of unwanted redness to 4=severe redness). The percentage of patients with at least a 1 grade decrease (improvement) on the SSA from baseline at Day 1 hour 1. Baseline was defined as the measurement at predose on Day 1.
Time Frame: Baseline, Day 1 (Hour 1)
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Pateints
Arm/Group | AGN-199201 | Vehicle
Number analyzed (Participants) | 222 | 218
Percentage of Pateints | 30.2 | 17.4

ADVERSE EVENTS:
Arm/Group | AGN-199201 | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/222 | 3/218
Other Adverse Events (participants affected / at risk) | 0/222 | 0/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-199201 (N=222) | Vehicle (N=218)
Fall (General disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1
Arteriosclerosis (Cardiac disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.